CLINICAL TRIAL: NCT03672305
Title: Single-center, Open Clinical Study on the Efficacy and Safety of c-Met/PD-L1 Chimeric Antigen Receptor T Cell Injection in the Treatment of Primary Hepatocellular Carcinoma
Brief Title: Clinical Study on the Efficacy and Safety of c-Met/PD-L1 CAR-T Cell Injection in the Treatment of HCC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, LiTao, Principal Investigator, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JGZNO1
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Primary Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- c-Met/PD-L1 CAR-T cells treating group (Other): Intervention Name:c-Met/PD-L1 CAR-T cell injection dosage form: injection dosage:The backtransfusion dose (recommended dose: 2 * 10^6/kg) was determined by the investigator based on the subject's own/disease condition and in vitro preparation.
  Interventions: Biological: c-Met/PD-L1 CAR-T cell injection

INTERVENTIONS:
Biological: c-Met/PD-L1 CAR-T cell injection — injection content:c-Met/PD-L1 CAR-T cell Infusion way:Steady intravenous drip in 15 to 30 minutes

SUMMARY:
Title: Single-center, open clinical study on the efficacy and safety of c-Met/PD-L1 T cell injection in the treatment of primary hepatocellular carcinoma

Stage: Phase I clinical trial

Purpose: To evaluate the efficacy and safety of c-Met/PD-L1 CAR-T cells in patients with primary hepatocellular carcinoma

Object: patients with primary hepatocellular carcinoma

Sample size: 50 cases

Number of centres：1

Study design: CT, MRI, PET and blood biochemical tests were performed before treatment to evaluate the state of HCC. Peripheral blood of the patient was extracted and PBMC was isolated. CAR-T cells were obtained by tranducing PBMC with c-Met/PD-L1 CAR lentivirus, and the proliferation capacity and immune phenotype of the cells were tested. After passing the inspection, the cells were re-injected into the patient three times. The efficacy and safety of c-Met/PD-L1 CAR-T cells was assessed respectively at 4 week, 12 week, 24 week and 48 week after treatment.

Trial product: c-Met/PD-L1 CAR-T cells

Course of treatment: 3 days for a course of treatment, only one course of treatment. A second course is given as appropriate if the treatment is beneficial to the patient.

DETAILED DESCRIPTION:
Title: Single-center, open clinical study on the efficacy and safety of c-Met/PD-L1 CAR-T cell injection in the treatment of primary hepatocellular carcinoma

Research purpose:

Primary outcome:

To evaluate the efficacy of c-Met/PD-L1 CAR-T cell injection in the treatment of primary hepatocellular carcinoma.

Secondary purpose:

1. To evaluate the clinical safety of c-Met/PD-L1 CAR-T cell injection in the treatment of primary hepatocellular carcinoma;
2. To assess the amplification and persistence of c-Met/PD-L1 CAR-T cells in subjects.

Study design:Single center, open clinical study

Subjects:Patients with primary hepatocellular carcinoma

Clinical trial cycle:

Screening stage:Selecting enrolled patients and collecting peripheral mononuclear cells; Treating stage: Pretreating and the backtransfusing c-Met/PD-L1 CAR-T cells Follow-up stage:Treatment was observed for 28 days (short-term follow-up), 28 days to 24 weeks (mid-term follow-up), and 24 weeks to progression/death (long-term follow-up);

Trial product:

Trial product:c-Met/PD-L1 CAR-T cells Dosage:The backtransfusion dose was determined by the investigator based on the subject's own/disease condition and in vitro preparation (recommended dose: 2 * 10^6/kg); Infusion way:Steady intravenous drip within 15 to 30 minutes

Clinical trial procedure:

1. The screening period:

   The subjects signed the informed consent form and performed a series of examinations according to the interview flow chart. The researchers judged whether the subjects met the inclusion criteria according to the examination results and inclusion/exclusion criteria, and did not meet the exclusion criteria. If the subjects were enrolled, peripheral blood mononuclear cells were collected, and the collection standard was 2-4 * 10^8 white blood cells;
2. nonmyeloablative pretreatment:(The following options are selected on a case-by-case basis)

   1. Fludarabine+Cyclophosphamide (FC)
   2. Bis-1-nitrosourea+Etoposide+Arabinoside+Cyclophosphamide (BECA);
3. Retransfusion period:

   The specific time and dose of retransfusion can be determined by the researchers;
4. Short-term follow-up period:

   Subjects will undergo a series of examinations according to the visit flow chart within 28 days after the expected dose of c-Met/PD-L1 CAR-T cells injection.The short-term efficacy and safety of c-Met/PD-L1 CAR-T cells injection were evaluated by the researchers based on the test results.
5. Mid-term follow-up:

   Subjects will undergo a series of examinations according to the visit flow chart 28 days to 24 weeks after re-transfusion of c-Met/PD-L1 CAR-T cells injection.The researchers will evaluate the mid-term efficacy and safety of c-Met/PD-L1 CAR-T cells based on the test results.
6. Long-term follow-up:

   Subjects will undergo a series of examinations according to the visit flow chart 24 weeks later until progress or death after retransfusion of c-Met/PD-L1 CAR-T cells.The long-term efficacy and safety of c-Met/PD-L1 CAR-T cells will be evaluated according to the test results.
7. Withdrawal visit (at any time) :All subjects may withdraw from this study at any stage of the trial.If the subjects withdraw from the study after returning to the c-Met/PD-L1 CAR-T cells, they shall complete the inspection items required in the visit flow chart, and the reason for the withdrawal shall be recorded in detail by the researchers.If the subject passes screening but withdraws from the visit before returning to the c-Met/PD-L1 CAR-T cells, only the baseline and screening tests need to be completed, and the reason for withdrawal will be recorded in detail by the investigators.If the subject withdraws from the screening test before the end of the screening test, only the screening test shall be completed and the reason for withdrawal shall be recorded in detail by the investigators.If treatment is discontinued due to adverse reactions (AE), the investigators will follow up with the necessary safety until the subjects return to baseline or to a stable state.

Evaluation index Main evaluation index

1. Objective tumor remission rate (ORR),complete remission (CR) and partial remission (PR) at 4 weeks, 12 weeks, 24 weeks and 48 weeks after treatment with c-Met/PD-L1 CAR-T cells;
2. Overall survival
3. Progression free survival
4. Event-free survival

Secondary evaluation index

1. Incidence of treatment-related adverse events (level 3 or level 4 adverse reactions, CTCAE V4.03 criteria). These included adverse events related to the treatment of c-Met/PD-L1 CAR-T cells, severe adverse events and clinically significant laboratory abnormalities;
2. The amplification level of c-Met/PD-L1 CAR-T cells in the subjects varied with time;
3. Duration of c-Met/PD-L1 CAR-T cells in the subjects;
4. The abatement features of hepatocellular carcinoma in subjects.

Statistical analysis SPSS18.0 was used for statistical analysis

1. The primary and secondary end points were analyzed by intentionality. The statistical analysis method of the end point was used to describe tumor ORR according to different follow-up time. Kaplan-meier method and survival curve were used to describe OS, PFS and EFS
2. The statistical analysis method of the secondary study endpoint was to describe the occurrence number and incidence of treatment-related adverse events, and to compare the difference of vital signs and laboratory indexes before and after treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 70 years (including 18 and 70 years);
2. Immune histochemistry detection was confirmed as c-met positive ; hepatocellular carcinoma, and the patient has no effective treatment at present
3. Liver tissue type: non-diffuse hepatocellular carcinoma, no extra hepatic metastasis or portal vein infiltration;
4. Cirrhosis of the liver: child-pugh A grade or child-pugh B grade, child-pugh-turcotte score <7;
5. Routine blood test: white blood cell count (WBC) or 3 * 10^9/L, lymphocyte percentage (LY) 15% or higher, hemoglobin (Hb), 90g/L or higher, prothrombin time (PT), international standardization ratio (INR) 1.7 or less, or prothrombin time (PT) extend the 4 s or less, lymphocyte acuity 0.8 * 10^9/L;
6. The main tissues and organs of the patients are functioning well (if the organs do not meet the following standards, but the researchers believe that the diseases themselves can be included):

   1. Hepatic and pancreatic functions: alanine aminotransferase/aspartate aminotransferase (ALT/AST) is 5 times of normal value, total bilirubin (TBiL) is 3.0mg/dL, albumin (ALB) is 35g/L, serum lipase is 1.5 times of normal value, and serum amylase is 1.5 times of normal value. Renal function: creatinine <2 ULN
   2. Lung function: indoor oxygen saturation greater than or equal to 95% (without oxygen inhalation)
   3. Cardiac function: LVEF is greater than or equal to 40%
   4. The absolute number of neutrophils is greater than or equal to 0.75 * 10^9/L, and platelets are greater than or equal to 50 * 10^9/L
7. ECOG score 0-1 or Karnofsky performance status (card score) (KPS) is greater than 60, and the expected survival time is greater than or equal to 12 weeks;
8. There are adequate venipuncture or venous sampling channels and no contraindications for lymphocyte separation;
9. No anti-tumor therapy, including chemotherapy, radiotherapy and immunotherapy (such as immunosuppressive drugs), was received within 4 weeks before enrollment, and the toxicity response of previous treatment was restored to level 1 or less (except for low-level toxicity such as hair loss);
10. Female subjects of reproductive age must have negative serum or urine pregnancy test during screening, and male and female patients agree to take effective contraceptive measures during the trial;
11. There were no other serious complications;
12. Voluntarily sign informed consent.

Exclusion Criteria:

1. Women during pregnancy (positive urine/blood pregnancy test) or lactation; A male or female who has a plan to conceive within the last 1 year; Effective contraceptive (condom or birth control pill, etc.) cannot be guaranteed for 1 year after enrollment;
2. The patients had uncontrollable infection within 4 weeks before enrollment. However, prophylactic antibiotics, antiviral and antifungal infection treatment are allowed; Active hepatitis b hepatitis c; People infected with human immunodeficiency virus (HIV);
3. Suffering from severe autoimmune disease or immunodeficiency disease;
4. The patient is allergic to large molecular biological drugs such as antibodies or cytokines;
5. The patient who has mentally ill;
6. The patient has substance abuse/addiction;
7. The patient who has a history of hepatocellular carcinoma;
8. Having severe peptic ulcer or bleeding;
9. A patient who receives an organ transplant or waits for one;
10. Patients requiring anticoagulation (e.g., warfarin or heparin);
11. Patients requiring long-term antiplatelet therapy (aspirin > 300 mg/d; Clopidogrel dose > 75 mg/d);
12. Organ failure patient:

    1. Cardiac function: grade 3 or above according to the New York heart association (NYHA) standard
    2. Liver function: C level above, according to child-pugh standard
    3. Chronic kidney disease (CKD) stage 4 or above; Renal insufficiency or above
    4. Lung function: severe respiratory failure, involving other organs
    5. Brain function: abnormal central nervous system or disturbance of consciousness;
13. Systemic use of hormones within 4 weeks before enrollment (use of prednisone 20mg/ d or less is allowed, except for inhaled hormones);
14. The patient participated in other clinical trials within 4 weeks before enrollment;
15. The patient has been treated with radiation for the past four weeks;
16. Investigators determined that the patient was unable or unwilling to comply with protocol requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
The efficacy of c-Met/PD-L1 CAR-T cells in the treatment of HCC | 6 months after treatment
  assessing the efficacy of c-Met/PD-L1 CAR-T cells through overall survival

SECONDARY OUTCOMES:
the incidence of treatment-emergent adverse events of c-Met/PD-L1 T cell injection in the treatment of HCC | 6 months after treatment
  the level 3 or level 4 adverse reactions according to CTCAE V4.03 standard
The amplification and persistence of c-Met/PD-L1 CAR-T cell in the subjects varied with time | 6 months after treatment
  The amplification level of c-Met/PD-L1 CAR-T cells varied with time and the duration of anti-c-met/pd-l1 CAR-T cells in the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Guozhong Ji, archiater, Study Chair — Second affiliated hospital of nanjing medical university

REFERENCES:
- [Background] Li YW, Yang FC, Lu HQ, Zhang JS. Hepatocellular carcinoma and hepatitis B surface protein. World J Gastroenterol. 2016 Feb 14;22(6):1943-52. doi: 10.3748/wjg.v22.i6.1943. PMID 26877602
- [Background] McGlynn KA, Petrick JL, London WT. Global epidemiology of hepatocellular carcinoma: an emphasis on demographic and regional variability. Clin Liver Dis. 2015 May;19(2):223-38. doi: 10.1016/j.cld.2015.01.001. Epub 2015 Feb 26. PMID 25921660
- [Background] Tagliamonte M, Petrizzo A, Tornesello ML, Ciliberto G, Buonaguro FM, Buonaguro L. Combinatorial immunotherapy strategies for hepatocellular carcinoma. Curr Opin Immunol. 2016 Apr;39:103-13. doi: 10.1016/j.coi.2016.01.005. Epub 2016 Feb 4. PMID 26851637
- [Background] Kenderian SS, Ruella M, Gill S, Kalos M. Chimeric antigen receptor T-cell therapy to target hematologic malignancies. Cancer Res. 2014 Nov 15;74(22):6383-9. doi: 10.1158/0008-5472.CAN-14-1530. Epub 2014 Nov 4. PMID 25371415
- [Background] Pico de Coana Y, Choudhury A, Kiessling R. Checkpoint blockade for cancer therapy: revitalizing a suppressed immune system. Trends Mol Med. 2015 Aug;21(8):482-91. doi: 10.1016/j.molmed.2015.05.005. Epub 2015 Jun 16. PMID 26091825
- [Background] Brentjens RJ, Riviere I, Park JH, Davila ML, Wang X, Stefanski J, Taylor C, Yeh R, Bartido S, Borquez-Ojeda O, Olszewska M, Bernal Y, Pegram H, Przybylowski M, Hollyman D, Usachenko Y, Pirraglia D, Hosey J, Santos E, Halton E, Maslak P, Scheinberg D, Jurcic J, Heaney M, Heller G, Frattini M, Sadelain M. Safety and persistence of adoptively transferred autologous CD19-targeted T cells in patients with relapsed or chemotherapy refractory B-cell leukemias. Blood. 2011 Nov 3;118(18):4817-28. doi: 10.1182/blood-2011-04-348540. Epub 2011 Aug 17. PMID 21849486
- [Background] Vesely MD, Kershaw MH, Schreiber RD, Smyth MJ. Natural innate and adaptive immunity to cancer. Annu Rev Immunol. 2011;29:235-71. doi: 10.1146/annurev-immunol-031210-101324. PMID 21219185
- [Background] Dotti G, Savoldo B, Brenner M. Fifteen years of gene therapy based on chimeric antigen receptors: "are we nearly there yet?". Hum Gene Ther. 2009 Nov;20(11):1229-39. doi: 10.1089/hum.2009.142. PMID 19702437
- [Background] Park TS, Rosenberg SA, Morgan RA. Treating cancer with genetically engineered T cells. Trends Biotechnol. 2011 Nov;29(11):550-7. doi: 10.1016/j.tibtech.2011.04.009. Epub 2011 Jun 12. PMID 21663987
- [Background] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Background] Davila ML, Riviere I, Wang X, Bartido S, Park J, Curran K, Chung SS, Stefanski J, Borquez-Ojeda O, Olszewska M, Qu J, Wasielewska T, He Q, Fink M, Shinglot H, Youssif M, Satter M, Wang Y, Hosey J, Quintanilla H, Halton E, Bernal Y, Bouhassira DC, Arcila ME, Gonen M, Roboz GJ, Maslak P, Douer D, Frattini MG, Giralt S, Sadelain M, Brentjens R. Efficacy and toxicity management of 19-28z CAR T cell therapy in B cell acute lymphoblastic leukemia. Sci Transl Med. 2014 Feb 19;6(224):224ra25. doi: 10.1126/scitranslmed.3008226. PMID 24553386
- [Background] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Background] Maus MV, Grupp SA, Porter DL, June CH. Antibody-modified T cells: CARs take the front seat for hematologic malignancies. Blood. 2014 Apr 24;123(17):2625-35. doi: 10.1182/blood-2013-11-492231. Epub 2014 Feb 27. PMID 24578504
- [Background] Maude SL, Barrett D, Teachey DT, Grupp SA. Managing cytokine release syndrome associated with novel T cell-engaging therapies. Cancer J. 2014 Mar-Apr;20(2):119-22. doi: 10.1097/PPO.0000000000000035. PMID 24667956
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Brudno JN, Kochenderfer JN. Toxicities of chimeric antigen receptor T cells: recognition and management. Blood. 2016 Jun 30;127(26):3321-30. doi: 10.1182/blood-2016-04-703751. Epub 2016 May 20. PMID 27207799